CLINICAL TRIAL: NCT00338234
Title: Observational Study of Iron Metabolism in Anemia in ICU and Post-Operative Patients, Role of Hepcidin
Brief Title: Observational Study of Iron Metabolism in Anemia in ICU and Post-Operative Patients
Acronym: FAIRe
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Société Française d'Anesthésie et de Réanimation (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sigismond LASOCKI, CHU BICHAT-Claude BERNARD
Other Study IDs: FAIRe
Record Dates: First submitted 2006-06-16; First posted 2006-06-20 (Estimated); Last update posted 2008-05-06 (Estimated); Status verified 2007-04

CONDITIONS: Anemia; Intensive Care; Cardiac Surgery
Keywords: anemia; intensive care; cardiac surgery; iron metabolism; hepcidin
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cardiac surgery: Successive cardiac surgery patients
- Surgical ICU: Successive patients admitted to the surgical ICU for more than 7 days, and experiencing anemia

SUMMARY:
Anemia in intensive care and post-operative patients is due to both blood loss (leading to iron loss) and inflammation.

DETAILED DESCRIPTION:
Anemia in intensive care and post-operative patients is due to both blood loss (leading to iron loss) and inflammation. The latter is known to interfere with iron metabolism, inducing iron storage instead of using it for hemoglobin synthesis. The discover of a new regulatory hormone of iron metabolism, hepcidin, may help us to better understand the link between inflammation and iron functional deficit. The aim of our study is to observe the variation of usual iron metabolism biological markers and of hepcidin, in order to define the better marker of iron loss in these clinical situations.

ELIGIBILITY:
Inclusion Criteria:

* Anemia (haemoglobin < 10 g/dL)
* Hospitalization in ICU for an expected duration of 7 days or more
* Or, day one post cardiac surgery

Exclusion Criteria:

* Chronic anemia (Hb < 9 g/dL for more than one month before hospitalization)
* Iron metabolism disease

Ages: 20 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * For the surgery :population 20 yers to 88 years old
  * For the reanimation : population to the 41 years to 85 years old
Sampling Method: Non-Probability Sample
Enrollment: 153 (Actual)
Dates: Start 2006-06; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Functional iron deficiency | during the study

SECONDARY OUTCOMES:
fatigue assessed by the MFI20 score for cardiac surgery patients | at one day,at seven days and at 28 days

CONTACTS AND LOCATIONS:
Overall Officials: sigismond lasocki, MD, Principal Investigator — Assistance Publique Hopitaux de Paris; Carole Beaumont, PhD, Study Chair — Institut National de la Santé Et de la Recherche Médicale, France; Isabelle Boutron, MD, Study Chair — Institut National de la Santé Et de la Recherche Médicale, France
Locations (1):
- APHP, hopital Bichat, Paris, France